CLINICAL TRIAL: NCT02173483
Title: Anterior Cruciate Ligament-reconstruction: Quadriceps Tendon or Hamstrings Tendon? A Prospective Randomised Controlled Trial
Brief Title: Anterior Cruciate Ligament-reconstruction: Quadriceps Tendon or Hamstrings Tendon? A Prospective Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Martin Lind, Professor, Aarhus University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: Danish EC - 110728514
Record Dates: First submitted 2014-06-17; First posted 2014-06-25 (Estimated); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Ligament; Laxity, Knee; Rupture of Anterior Cruciate Ligament
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Quadriceps graft (Other): Proximally from patella the Quadriceps graft is harvested and used as a knew anterior cruciate ligament after rupture.
  Interventions: Procedure: Quadriceps graft
- Hamstrings Graft (Other): The Hamstrings graft is harvested and used as a knew anterior cruciate ligament after rupture.
  Interventions: Procedure: Quadriceps graft

INTERVENTIONS:
Procedure: Quadriceps graft

SUMMARY:
The purpose of this study is to determine whether there is a difference in muscle strength after anterior cruciate ligament comparing 2 surgery technics. Using either autograft hamstrings tendon or a autograft quadriceps tendon.

ELIGIBILITY:
Inclusion Criteria:

* Anterior cruciate ligament rupture

Exclusion Criteria:

* current malignant disease
* Rheumatoid arthritis
* Other knee ligament instability
* Obesity BMI >30
* Morbus Bechterew

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-05; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Patient reported outcome score - IKDC | 12 month
  IKDC (international Knee Documentation committee) subjective score (0-100)

SECONDARY OUTCOMES:
Knee laxity | 12 month
  KT-1000 arthrometer
Patient reported outcome score - KOOS | 12 month
  Koos (Knee injury and Osteoarthritis Outcome Score) contains 5 subscores (Pain, ADL, QOL, Symptoms, Sport & recreation). Each subscore ranges from 0-100 where higher values represent a better score.
TEGNER | 12 month
  Patient reported outcome score (range 0-10)
Anterior knee pain scale | 12 month
  Patient reported outcome score (range 0-100)
Donor Site morbidity score | 12 month
  Patient reported outcome score (range 100-0)

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Sports Trauma, Tage-Hansens Gade 2b, Aarhus, Denmark

REFERENCES:
- [Derived] Sinding KS, Nielsen TG, Hvid LG, Lind M, Dalgas U. Effects of Autograft Types on Muscle Strength and Functional Capacity in Patients Having Anterior Cruciate Ligament Reconstruction: A Randomized Controlled Trial. Sports Med. 2020 Jul;50(7):1393-1403. doi: 10.1007/s40279-020-01276-x. PMID 32125668
- [Derived] Lind M, Nielsen TG, Soerensen OG, Mygind-Klavsen B, Fauno P. Quadriceps tendon grafts does not cause patients to have inferior subjective outcome after anterior cruciate ligament (ACL) reconstruction than do hamstring grafts: a 2-year prospective randomised controlled trial. Br J Sports Med. 2020 Feb;54(3):183-187. doi: 10.1136/bjsports-2019-101000. Epub 2019 Nov 8. PMID 31704697